CLINICAL TRIAL: NCT06043544
Title: Hymovis® Intra-articular Injections vs Corticosteroids Intra-articular Injections in Patients Affected by Glenohumeral Osteoarthritis: a Monocentric Randomized Open-label Trial
Brief Title: Hymovis® Intra-articular Injections vs Corticosteroids Intra-articular Injections in Patients Affected by Glenohumeral Osteoarthritis:
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Concordia Hospital Rome (Other)
Responsible Party: Principal Investigator, Nicola de Gasperis, Principal Investigator, Concordia Hospital Rome
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hymovis 10-04-21
Record Dates: First submitted 2023-08-29; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Glenohumeral Osteoarthritis
Keywords: Osteoarthritis; Hyaluronic Acid; Corticosteroids
MeSH Terms: conditions — Osteoarthritis | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Intervention Model Description: 80 consecutive patients with glenohumeral OA degree II or III were prospectively enrolled in our clinic from May 2021 to March 2022. The study was approved by Concordia Hospital Ethical Committee (02/2021) and performed according to ISO14155:2020 and Declaration of Helsinki.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Experimental): patients shoulder treated with Hymovis® 24mg/3ml.
  Interventions: Device: Hyaluronic Acid 24 MG in 3 mL Prefilled Syringe
- Control group (Active Comparator): patients shoulder treated with Corticosteroid.
  Interventions: Drug: Corticosteroid injection

INTERVENTIONS:
Device: Hyaluronic Acid 24 MG in 3 mL Prefilled Syringe — Patients in the treatment group received two intra-articular injections with Hymovis® (24mg/3ml) a week apart from each other
  Arms: Treatment group
Drug: Corticosteroid injection — Patients in control group received two intra-articular injections with corticosteroids a week apart from each other.
  Arms: Control group

SUMMARY:
This monocentric randomized open-label study aims to assess the efficacy and safety of a treatment with medium molecular weight hyaluronic acid (HA) compared to a treatment with corticosteroids on patients affected by glenohumeral osteoarthritis.

DETAILED DESCRIPTION:
Glenohumeral osteoarthritis (OA) is a very common joint disease characterized by pain and functional limitation. No standardized protocols of treatment are available in clinical practice and literature data are confusing. This monocentric randomized open-label study aims to assess the efficacy and safety of a treatment with medium molecular weight hyaluronic acid (HA) compared to a treatment with corticosteroids on patients affected by glenohumeral osteoarthritis.

A total of 80 consecutive patients with glenohumeral OA (Kellegren Lawrence degree II or III) were randomized in two different groups, intto Hymovis® (24mg/3ml) (treatment group) or into corticosteroids (control group), with a follow-up after 3 and 6 months. Modifications in terms of pain (VAS), range of motion (ROM) and quality of life (EQ-5D) were observed during the treatment.

ELIGIBILITY:
Inclusion Criteria:

Male or female patient aged ≥40 years

Patient suffering from glenohumeral osteoarthritis with chronic shoulder pain. Chronic shoulder pain is defined as follows:

* Persistence for a period of at least 6 months, but not more than 5 years;
* Pain perceived by the patient with a frequency of at least 50% of the days in the month preceding the inclusion visit; Kellgren-Lawrence grade of 2 or 3 in the glenohumeral joint confirmed by x-ray exam performed within 3 months prior to the inclusion visit.

Presence, at baseline, of pain on movement, in the shoulder under study, measured by VAS with a score between 40 and 80 mm Presence at baseline of pain in the contralateral shoulder at least 10mm less than the study shoulder and no more than 40mm as measured by VAS at the inclusion visit

Presence, at baseline, of limitation of shoulder motion in at least one direction in the following ranges of motion:

* Fixed scapula abduction ≤ 80°
* Internal rotation in abduction ≤ 55°
* External rotation in abduction ≤ 80° These shoulder limitations are for normal expected excursions. Patient who has not responded adequately to non-pharmacological conservative therapy and to taking simple analgesics Patient willing to sign and able to understand the Informed Consent form Patient who is not pregnant or nursing. Women of childbearing potential (including women who have been less than one year postmenopausal) must agree to use reliable contraception for the duration of the study.

Exclusion Criteria:

* Presence, on clinical evaluation, of adhesive capsulitis
* Evidence of rotator cuff injury
* Presence of primary extra-articular shoulder syndromes (eg impingement, bursitis, tendonitis)
* Evidence of clinically significant shoulder deformity
* Signs, evident on X-ray radiography of the shoulder, of recent fractures, severe loss of bone density and/or severe deformity
* Diagnosed with crystal deposition disease of calcium pyrophosphate dihydrate (CPPD) or chondrocalcinosis of the shoulder
* Presence of pathology of the cervical vertebrae (able to alter the clinical evaluation) which, in the three months preceding the inclusion visit, was symptomatic and required active treatment
* Presence of any active musculoskeletal disease affecting the diagnosis/evaluation of shoulder pain or presence of pain of any neurological etiology and acute shoulder infection
* Presence of major surgery, arthroplasty or arthroscopy in the shoulder under study in the 6 months prior to inclusion and/or surgery planned during the study
* Patient undergoing local radiotherapy for breast cancer
* Patient with polymyalgia rheumatica
* History of skin cancer (except basal cell carcinoma) treated for less than two years
* History of severe recurrent or immune-mediated allergic reactions
* Presence of infection and/or skin pathologies in the injection area; psoriasis
* Presence of serious gastrointestinal, renal, hepatic, pulmonary, cardiovascular, neurological disorders that could interfere with the study results or patient's inability to comply with the study requirements
* Known allergy or suspected allergic reactions to hyaluronate or corticosteroid preparations
* Taking HA products intra-articularly in the month preceding the inclusion visit
* Taking bisphosphonates and/or pharmaceutical products taken orally and containing glucosamine and/or chondroitin sulphate and/or diacerin (eg Chondrosulf, Structum 500, Dona, Viatril, Fisiodar, Artrodar, etc.) in the month preceding the inclusion visit unless the dosage was stable in the two months prior to the inclusion visit
* Intra-articular corticosteroid injections in the study shoulder in the three months preceding the inclusion visit
* Intra-articular corticosteroid injections in any joint in the month preceding the inclusion
* Taking oral corticosteroids in the month prior to the inclusion visit (only inhaled corticosteroids are permitted)
* Previous use of HA in the study shoulder within 6 months prior to inclusion
* Changed physical therapy in the month prior to inclusion visit or unwillingness to maintain stable regimen
* Patient with history of thyroid insufficiency
* Patient being treated with anticoagulant therapy
* Patient on phenobarbital treatment prior to study inclusion
* Taking analgesic therapies (NSAIDs, opioid analgesics, topical analgesics) for any condition that could interfere with the evaluation of the shoulder under study
* Intake of another experimental product in the month preceding the inclusion visit
* Patient who, in the opinion of the investigator, is unwilling to comply with study procedures or will not cooperate during the course of the study
* Pregnant or breastfeeding woman

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-05-02 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Evaluate the pain reduction in the target shoulder compared to control group | At 6 months
  Changes of pain on movement in the target shoulder, evaluated with a 0-100 mm Visual Analogue Scale (VAS) values compared to baseline (V1).

SECONDARY OUTCOMES:
Evaluation of the Quality of Life of the patients | At 6 months
  Changes of patient's quality of life, evaluated by administration of the EuroQol 5-Dimension Questionnaire (EQ-5D-5L) compared to baseline (V1)
Evaluate the amelioration of shoulder functionality | At 6 months
  Clinical functional assessment on movement from baseline (V1), measured by Constant Murley (CMS) shoulder test ;
Evaluate the pain reduction in the target shoulder compared to baseline | At 6 months
  Changes of pain on movement in the target shoulder, evaluated with a 0-100 mm Visual Analogue Scale (VAS) values compared to baseline (V1).
Evaluation of the safety of the treatment | 12 months
  Safety of Hymovis® were evaluated in terms of incidence of treatment-emergent adverse events (TEAEs) over the investigational period.

CONTACTS AND LOCATIONS:
Locations (1):
- Concordia Hospital, Rome, Italy